CLINICAL TRIAL: NCT02402218
Title: CHAMPS Study: Chronic HepAtitis C Management to ImProve OutcomeS
Acronym: CHAMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00055591; 5R01DA016065-12 (NIH)
Record Dates: First submitted 2015-03-18; First posted 2015-03-30 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Hepatitis C Virus Infection, Response to Therapy of; Human Immunodeficiency Virus
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (Active Comparator): Participants receive standard of care for Hepatitis C in the clinic.
  Interventions: Other: Usual Care
- Usual care plus peer-mentors (Experimental): In addition to receiving standard of care for HCV in the clinic, this is an investigational strategy in which participants assigned to this group will be asked to interact with a peer-mentor who is someone who has been cured of their HCV infection.
  Interventions: Other: Usual care plus peer-mentors
- Usual care plus incentives (Experimental): In addition to receiving standard of care for HCV in the clinic, this is an investigational strategy in which participants assigned to this group will be given incentives after completing certain goals during the course of the study.
  Interventions: Other: Usual care plus incentives

INTERVENTIONS:
Other: Usual care plus peer-mentors — Participants are assigned a peer mentor for support before and after treatment for HCV with Harvoni.
  Arms: Usual care plus peer-mentors
Other: Usual care plus incentives — Participants are given incentives after completing treatment goals.
  Arms: Usual care plus incentives
Other: Usual Care — Participants receive standard of care in the clinic from their health care team.
  Arms: Usual Care

SUMMARY:
This study is being done to compare three strategies to deliver HCV treatment with ledipasvir/sofosbuvir which is an approved therapy which is administered as one tablet by mouth daily for 12 weeks. The study population is persons living with HIV and hepatitis C virus (HCV) coinfection who also use drugs. Participants will be randomized into one of three treatment groups:

1. Usual care in the clinic. This treatment group will receive the standard of care for HCV treatment from their health care team.
2. Usual care plus peer-mentors. In addition to the usual care, this is an investigational strategy in which participants assigned to this group will be asked to interact with a peer-mentor who is someone who has been cured of their HCV infection.
3. Usual care plus incentives. In addition to the usual care, this is an investigational strategy in which participants assigned to this group will be given incentives after completing certain treatment goals during the course of the study.

HCV treatment with ledipasvir/sofosbuvir is considered the standard of care for HCV and is recommended by experts in liver disease and infectious diseases.

DETAILED DESCRIPTION:
Recent advances in Hepatitis C Virus (HCV) treatment represent a paradigm shift for the treatment of HCV-infected persons with Human Immunodeficiency Virus (HIV) coinfection. With potent antiviral activity, excellent safety/tolerability, few drug interactions and once daily, oral dosing, Sofosbuvir (SOF)/Ledipasvir (LDV) have had excellent efficacy in randomized controlled trials and offer great promise for the treatment of hepatitis C in HIV/HCV coinfected patients who are at high risk for progressive liver disease and HCV-related mortality. While the availability of SOF/LDV has great promise for the treatment of patients, the experience with antiretroviral therapy (ART) for the treatment of HIV infection indicates that interferon-free oral therapy is necessary but not sufficient to cure HCV in the real world. While removal of Interferon increases the proportion of coinfected persons who use drugs (PWUD) eligible for treatment, multiple barriers will remain (e.g., medical/psychiatric illness, substance abuse, and social constraints). Effective ART in coinfected PWUDs provides a strategic framework for the delivery of curative HCV treatment; novel and effective strategies for delivering this care for HCV must be evaluated, including incentives and peer-mentoring.

Financial incentives. One method for increasing delivery of care is the contingent administration of monetary incentives; such reinforcements have improved health outcomes related to drug/alcohol abstinence, smoking cessation, childhood vaccination, tuberculosis care and HIV treatment. Contingent reinforcement has also been successfully used to link HIV-infected patients to care and improve adherence to ART. Curative HCV treatments are given for a finite duration (12 weeks) which offers an ideal paradigm for incentive interventions by reducing the overall cost and removing concerns of loss of adherence if incentives are stopped.

Peer support. A second method for improving delivery of care is the use of peers or laypersons with the same illness. By matching on cultural competencies and establishing trust, peers may be particularly effective in some settings. In one study, African American veterans with poorly controlled diabetes assigned to peer-support had better glucose control than those assigned financial incentives. Coinfected patients may benefit from peer support.

The investigators will test two innovative strategies to improve HCV treatment outcomes in HIV/HCV coinfected patients through the delivery of SOF/LDV for 12 weeks as part of a randomized controlled trial. HIV-infected patients will receive SOF/LDV under one of three randomly assigned conditions: usual care (clinic-based nursing model), incentive care (IC) or peer-mentor care (PMC).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or greater
* Hepatitis C genotype 1 infection for at least 6 months
* No evidence of Hepatocellular Carcinoma or End-Stage Liver Disease (e.g., history of ascites, bleeding varices, and/or encephalopathy)
* Cluster of Differentiation 4 (CD4) cell count > 100 cells/mm3 for more than 3 months
* HIV RNA positive for more than 3 months
* Ability to communicate effectively with key study personnel
* Willing to give written informed consent and comply with the study requirements
* Life expectancy > 2 year

Exclusion Criteria:

* Currently receiving Hepatitis C treatment
* Renal insufficiency - estimated glomerular filtration rate, calculated by the chronic kidney disease epidemiology collaboration formula: <30 mL/min/1.73 m2
* Antiretroviral therapy inclusive of STRIBILD or APTIVUS
* Inability or unwillingness to avoid pregnancy for woman of child-bearing potential and/or to father children during treatment and for a period of 3 months following completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sulkowski, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hospital : The John G. Bartlett Specialty Practice, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ward KM, Falade-Nwulia O, Moon J, Sutcliffe CG, Brinkley S, Haselhuhn T, Katz S, Herne K, Arteaga L, Mehta SH, Latkin C, Brooner RK, Sulkowski MS. A Randomized Controlled Trial of Cash Incentives or Peer Support to Increase HCV Treatment for Persons With HIV Who Use Drugs: The CHAMPS Study. Open Forum Infect Dis. 2019 Apr 9;6(4):ofz166. doi: 10.1093/ofid/ofz166. eCollection 2019 Apr. PMID 31049365

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between August 2015 and October 2016 at an outpatient clinic in Baltimore, MD, USA.
Groups:
- Usual Care Plus Peer-mentors: In addition to receiving standard of care for hepatitis C virus (HCV) in the clinic, this is an investigational strategy in which participants assigned to this group will be asked to interact with a peer-mentor who is someone who has been cured of their HCV infection.
  Usual care plus peer-mentors: Participants are assigned a peer mentor for support before and after treatment for HCV with Harvoni.
Period: Overall Study
Arm/Group | Usual Care | Usual Care Plus Peer-mentors | Usual Care Plus Incentives
Started | 36 | 54 | 54
Initiated Treatment With LDV/SOF | 24 | 45 | 41
Completed Treatment With LDV/SOF | 23 | 42 | 39
Achieved Sustained Virologic Response | 22 | 41 | 37
Completed | 22 | 41 | 37
Not Completed | 14 | 13 | 17
Not completed — Did not pickup study medication | 12 | 9 | 13
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Reinfection | 0 | 0 | 1
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Usual Care Plus Peer-mentors | Usual Care Plus Incentives | Total
Number analyzed (Participants) | 36 | 54 | 54 | 144
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55.8 [51.8 to 60.2] | 55.1 [50.5 to 59.3] | 54.0 [48.8 to 59.2] | 54.9 [50.6 to 59.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 19 | 23 | 56
  Male | 22 | 35 | 31 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 36 | 54 | 54 | 144
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 33 | 52 | 48 | 133
  White | 3 | 2 | 6 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 54 | 54 | 144
Marital Status [Count of Participants; unit: Participants]
  Never Married | 19 | 27 | 26 | 72
  Married | 5 | 13 | 5 | 23
  Separated | 3 | 3 | 5 | 11
  Divorced | 6 | 8 | 9 | 23
  Widowed | 3 | 3 | 9 | 15
Employment Status [Count of Participants; unit: Participants]
  Employed | 6 | 7 | 9 | 22
  Unemployed | 30 | 47 | 45 | 122
Has Health Insurance [Count of Participants; unit: Participants]
  Has Health Insurance | 36 | 54 | 54 | 144
  Does Not Have Health Insurance | 0 | 0 | 0 | 0
Substance Use History- Self Report [Count of Participants; unit: Participants]
  Self-report use of cocaine or heroin- lifetime: Yes | 35 | 48 | 48 | 131
  Self-report use of cocaine or heroin- lifetime: No | 1 | 6 | 6 | 13
  Self-report use of cocaine or heroin- last 30 days: Yes | 12 | 12 | 12 | 36
  Self-report use of cocaine or heroin- last 30 days: No | 24 | 42 | 42 | 108
  Self-Report of Drug Use (any) in the Last 2 Years: Yes | 24 | 33 | 33 | 90
  Self-Report of Drug Use (any) in the Last 2 Years: No | 12 | 21 | 21 | 54
Urine Toxicology [Count of Participants; unit: Participants] — Population: 5 participants in the usual care group and 3 participants in the peer mentor group did not complete a urine toxicology at baseline.
  Participants
    Not Done: number analyzed (Participants) | 31 | 51 | 54 | 136
    Not Done | 5 | 3 | 0 | 8
    Benzodiazepine: number analyzed (Participants) | 31 | 51 | 54 | 136
    Benzodiazepine | 3 | 5 | 6 | 14
    Cocaine: number analyzed (Participants) | 31 | 51 | 54 | 136
    Cocaine | 12 | 12 | 19 | 43
    Heroin: number analyzed (Participants) | 31 | 51 | 54 | 136
    Heroin | 6 | 16 | 14 | 36
    Cannabinoid: number analyzed (Participants) | 31 | 51 | 54 | 136
    Cannabinoid | 9 | 19 | 13 | 41
    Methadone: number analyzed (Participants) | 31 | 51 | 54 | 136
    Methadone | 10 | 15 | 13 | 38
    Oxycod/ Oxymorph: number analyzed (Participants) | 31 | 51 | 54 | 136
    Oxycod/ Oxymorph | 4 | 1 | 4 | 9
    None of the Above Detected: number analyzed (Participants) | 31 | 51 | 54 | 136
    None of the Above Detected | 7 | 13 | 16 | 36
    Negative or only methadone: number analyzed (Participants) | 31 | 51 | 54 | 136
    Negative or only methadone | 10 | 16 | 19 | 45
    Negative or only methadone or oxycodone: number analyzed (Participants) | 31 | 51 | 54 | 136
    Negative or only methadone or oxycodone | 11 | 17 | 20 | 48
    Negative or only methadone or oxycodone or benzodi: number analyzed (Participants) | 31 | 51 | 54 | 136
    Negative or only methadone or oxycodone or benzodi | 11 | 18 | 23 | 52
    Negative or only methadone or oxycodone or marijua: number analyzed (Participants) | 31 | 51 | 54 | 136
    Negative or only methadone or oxycodone or marijua | 17 | 27 | 24 | 68
    Positive for cocaine only: number analyzed (Participants) | 31 | 51 | 54 | 136
    Positive for cocaine only | 1 | 3 | 4 | 8
    Positive for Heroin only: number analyzed (Participants) | 31 | 51 | 54 | 136
    Positive for Heroin only | 1 | 2 | 4 | 7
    Positive for cocaine and heroin only: number analyzed (Participants) | 31 | 51 | 54 | 136
    Positive for cocaine and heroin only | 1 | 2 | 1 | 4
    Positive for cocaine OR heroin: number analyzed (Participants) | 31 | 51 | 54 | 136
    Positive for cocaine OR heroin | 13 | 23 | 27 | 63
phosphatidylethanol (ng/mL) [Count of Participants; unit: Participants] — Population: 3 participants in the usual care group, 2 participants in the peer mentor group and 4 participants in the incentive care group did not complete a phosphatidylethanol test at baseline.
  Participants
    number analyzed (Participants) | 33 | 52 | 50 | 135
    <50 ng/mL | 18 | 33 | 37 | 88
    ≥50 ng/mL | 15 | 19 | 13 | 47
Self-report current alcohol use [Count of Participants; unit: Participants]
  Never | 14 | 23 | 22 | 59
  Monthly or Less | 9 | 12 | 12 | 33
  2-4x per month | 5 | 12 | 7 | 24
  2-3x per week | 5 | 4 | 5 | 14
  ≥4x per week | 3 | 3 | 8 | 14
alcohol use disorders identification test (AUDIT) [Count of Participants; unit: Participants] — The Alcohol Use Disorders Identification Test (AUDIT) was developed by the World Health Organization and includes 10 questions that assess alcohol use and drinking behaviors. For this study, AUDIT scores ≥8 for men and ≥4 for women were categorized as hazardous drinking. Scores range from 0 to 40, with higher scores indicating greater alcohol dependence.
  Participants
    Male <8 | 20 | 28 | 22 | 70
    Male ≥8 | 2 | 7 | 9 | 18
    Female <4 | 7 | 13 | 16 | 36
    Female ≥4 | 7 | 6 | 7 | 20
alcohol use disorders identification test (AUDIT) [Count of Participants; unit: Participants] — The Alcohol Use Disorders Identification Test (AUDIT) was developed by the World Health Organization and includes 10 questions that assess alcohol use and drinking behaviors. For this study, AUDIT scores ≥4 were categorized as hazardous drinking. Scores range from 0 to 40, with higher scores indicating greater alcohol dependence.
  Participants
    0-3 | 19 | 34 | 35 | 88
    4-7 | 13 | 10 | 8 | 31
    8-11 | 4 | 6 | 1 | 11
    ≥12 | 0 | 4 | 10 | 14
HIV RNA copies [Count of Participants; unit: Participants]
  ≤50 | 30 | 43 | 42 | 115
  >50 | 6 | 11 | 12 | 29
HIV RNA if ≥50 copies/mL [Median (Full Range); unit: copies/mL] | 20767 [251 to 101942] | 645 [55 to 357083] | 15903 [52 to 114561] | 5702 [52 to 357083]
Alanine Aminotransferase [Median (Full Range); unit: U/L] — Population: ALT not done for 1 participant in peer mentor group
  U/L
    number analyzed (Participants) | 36 | 53 | 54 | 143
    (all) | 39 [26 to 60] | 33 [20 to 46] | 29 [21 to 44] | 33 [21 to 50]
Aspartate Aminotransferase [Median (Full Range); unit: U/L] — Population: AST not done for 2 participants in peer group and 3 participants in incentive group
  U/L
    number analyzed (Participants) | 36 | 52 | 51 | 139
    (all) | 45 [34 to 60] | 39 [27 to 59] | 36 [30 to 59] | 40 [31 to 59]
Patient taking antiretroviral therapy [Count of Participants; unit: Participants]
  Yes | 35 | 52 | 52 | 139
  No | 1 | 2 | 2 | 5
HIV antiretroviral therapy (ART) Changed Pre-Treatment with Harvoni [Count of Participants; unit: Participants] — Population: This baseline measure only applies to the n=129 participants that saw a provider after enrollment in the study.
  Participants
    number analyzed (Participants) | 31 | 50 | 48 | 129
    Yes | 10 | 11 | 7 | 28
    No | 21 | 39 | 41 | 101
HCV Genotype/Subtype [Count of Participants; unit: Participants]
  1A | 29 | 40 | 43 | 112
  1B | 7 | 14 | 11 | 32
HCV RNA [Median (Full Range); unit: IU/mL] | 2730000 [472000 to 5740000] | 4790000 [1680000 to 10300000] | 2730000 [624000 to 8350000] | 2975000 [869000 to 8825000]
Liver Disease Stage by FibroScan [Median (Inter-Quartile Range); unit: kPa] — Population: 7 unsuccessful FibroScan measurements due to participant's body type
  kPa
    number analyzed (Participants) | 35 | 52 | 50 | 137
    (all) | 7.8 [5.4 to 9.9] | 6.8 [5.2 to 9.1] | 6.7 [5.1 to 8.6] | 6.9 [5.2 to 9.0]
Liver Disease Stage by FibroScan [Count of Participants; unit: Participants]
  ≤8 kPa | 20 | 34 | 36 | 90
  8.1-11.9 kPa | 11 | 13 | 7 | 31
  ≥12 kPa | 4 | 5 | 7 | 16
  Unsuccessful | 1 | 2 | 4 | 7
Cluster of differentiation 4 (CD4) Count [Median (Inter-Quartile Range); unit: cells/mm^3] | 453 [325 to 760] | 581 [387 to 851] | 509 [343 to 756] | 530 [340 to 797]
Centers for Depression Epidemiology Scale (CES-D) [Count of Participants; unit: Participants] — In this study, active depression is defined as score ≥16. This is a measure that asks patients to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
  Participants
    <16 | 16 | 20 | 20 | 56
    ≥16 | 20 | 34 | 34 | 88
Centers for Depression Epidemiology Scale (CES-D) [Count of Participants; unit: Participants] — Measure Description: In this study, severe active depression is defined as score ≥21. This is a measure that asks patients to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
  Participants
    <21 | 22 | 29 | 31 | 82
    ≥21 | 14 | 25 | 23 | 62
Number of times rescheduled or missed week 0 clinical appointment for initial evaluation [Count of Participants; unit: Participants]
  0 | 26 | 39 | 35 | 100
  1-2 | 9 | 10 | 16 | 35
  3+ | 1 | 5 | 3 | 9
Emotional Support [Count of Participants; unit: Participants] — Patient-Reported Outcomes Measurement Information System Short Form v2.0, Emotional Support 8a; low support defined as short form score <33
  Participants
    <33 | 11 | 24 | 21 | 56
    ≥33 | 25 | 30 | 33 | 88
Self-report fatigue [Count of Participants; unit: Participants] — Patient-Reported Outcomes Measurement Information System v1.0, Fatigue Short Form 7a; Fatigue defined as ≥16
  Participants
    <16 | 18 | 24 | 22 | 64
    ≥16 | 18 | 30 | 32 | 80
Primary Care Visit in the last 12 months [Count of Participants; unit: Participants] — Population: Self-report baseline measure not collected for 2 participants in the peer mentor group and 1 participant in the incentive care group.
  Participants
    number analyzed (Participants) | 36 | 52 | 53 | 141
    Yes | 36 | 48 | 52 | 136
    No | 0 | 4 | 1 | 5
Self-report "Do you think your doctor understands the pressure you are under outside of the clinic?" [Count of Participants; unit: Participants] — Population: Self-report baseline measure not collected for 2 participants in the peer mentor group and 1 participant in the incentive care group.
  Participants
    number analyzed (Participants) | 36 | 52 | 53 | 141
    Yes | 6 | 7 | 9 | 22
    No | 29 | 42 | 41 | 112
    Under No Pressure | 1 | 2 | 2 | 5
    Don't Know | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Initiated HCV Therapy by Intervention Group
Description: The percentage of participants who initiated HCV therapy [Ledipasvir/Sofosbuvir (LDV/SOF)] with Usual Care (UC), Incentive Care (IC), and Peer-Mentor Care (PMC).
Time Frame: at week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care Plus Peer-mentors | Usual Care Plus Incentives
Number analyzed (Participants) | 36 | 54 | 54
Participants | 24 | 45 | 41
Statistical Analysis 1: Comparison: Usual Care vs Usual Care Plus Peer-mentors vs Usual Care Plus Incentives; Sample size was based on an estimated HCV treatment initiation rate of 50% in the UC group (based on a 33% rate observed during the interferon era) and 80% in the intervention groups, a significance level of 0.05, a desired ratio of participants in the intervention group compared to UC group of 3 to 2, and power of 80% to detect this difference between groups. The study was not powered to detect differences between the peer and cash groups; Test type: Superiority; p = .11, Chi-squared — For the primary and secondary outcomes, the proportion of participants with the outcome in each group was compared using a chi-square test

2. Secondary Outcome: Sustained Virologic Response (SVR) Following Treatment by Intervention Group
Description: The number of participants who achieved SVR, defined as HCV RNA not detected at 12 weeks after completion of the HCV treatment regimen
Time Frame: at post-treatment week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care Plus Peer-mentors | Usual Care Plus Incentives
Number analyzed (Participants) | 36 | 54 | 54
Participants | 22 | 41 | 37
Statistical Analysis 1: Comparison: Usual Care vs Usual Care Plus Peer-mentors vs Usual Care Plus Incentives; Test type: Superiority; p = .22, Chi-squared

3. Secondary Outcome: Number of Participants With Adverse Events During HCV Treatment by Intervention Group
Description: Number of Participants who self-reported Adverse Events During HCV Treatment by Intervention Group
Time Frame: at post-treatment week 12
Population: Among participants that initiated treatment only.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care Plus Peer-mentors | Usual Care Plus Incentives
Number analyzed (Participants) | 24 | 45 | 41
Participants | 13 | 24 | 20

4. Secondary Outcome: Change in Alcohol Use by Blood Test During HCV Treatment
Description: Alcohol intake during HCV treatment measured using dried whole blood spots to measure the level of phosphatidylethanol (PEth) at pre-treatment and treatment week 6
Time Frame: Pre-treatment and at treatment week 6
Population: Participants that completed PEth tests at enrollment and week 6 of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care Plus Peer-mentors | Usual Care Plus Incentives
Number analyzed (Participants) | 22 | 41 | 35
Participants
  No change in alcohol use from week 0 to week 6 | 20 | 38 | 32
  Increase in alcohol use from week 0 to week 6 | 0 | 0 | 2
  Decrease in alcohol use from week 0 to week 6 | 2 | 3 | 1
Statistical Analysis 1: Comparison: Usual Care vs Usual Care Plus Peer-mentors vs Usual Care Plus Incentives; changes in the frequency of drug and alcohol use before and during treatment were compared using chi-square tests to evaluate the safety of cash incentives; Test type: Superiority; p = 0.33, Chi-squared

5. Secondary Outcome: Change in Illicit Drug Use During HCV Treatment
Description: Illicit drug use during HCV treatment measured by urine toxicology testing pre-treatment and at treatment week 6
Time Frame: Pre-treatment and at treatment week 6
Population: Participants that completed urine toxicology tests at enrollment and week 6 of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care Plus Peer-mentors | Usual Care Plus Incentives
Number analyzed (Participants) | 24 | 45 | 41
Participants
  No change in cocaine or heroin use from wk 0 to 6 | 16 | 37 | 34
  Increase in cocaine or heroin use from wk 0 to 6 | 5 | 4 | 2
  Decrease in cocaine or heroin use from wk 0 to 6 | 3 | 4 | 5
Statistical Analysis 1: Comparison: Usual Care vs Usual Care Plus Peer-mentors vs Usual Care Plus Incentives; Test type: Superiority; p = 0.30, Chi-squared — changes in the frequency of drug and alcohol use before and during treatment were compared using chi-square tests to evaluate the safety of cash incentives

6. Secondary Outcome: Number of Participants With Re-Infection After Achieving Sustained Virologic Response by Intervention Group
Description: Number of persons who achieved sustained virologic response following treatment who subsequently have HCV RNA detected with a new strain of the virus.
Time Frame: at post-treatment week 12
Population: Among participants that initiated treatment only.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Usual Care Plus Peer-mentors | Usual Care Plus Incentives
Number analyzed (Participants) | 24 | 45 | 41
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From treatment initiation to post-treatment week 12
Groups:
- Usual Care With LDV/SOF: Participants receive standard of care for Hepatitis C in the clinic.
  Usual Care: Participants receive standard of care in the clinic from their health care team. This group of patients initiated treatment with LDV/SOF.
- Usual Care Plus Peer-mentors With LDV/SOF: In addition to receiving standard of care for HCV in the clinic, this is an investigational strategy in which participants assigned to this group will be asked to interact with a peer-mentor who is someone who has been cured of their HCV infection.
  Usual care plus peer-mentors: Participants are assigned a peer mentor for support before and after treatment for HCV with LDV/SOF. This group of patients initiated treatment with LDV/SOF.
- Usual Care Plus Incentives With LDV/SOF: In addition to receiving standard of care for HCV in the clinic, this is an investigational strategy in which participants assigned to this group will be given incentives after completing certain goals during the course of the study.
  Usual care plus incentives: Participants are given incentives after completing treatment goals. This group of patients initiated treatment with LDV/SOF.
Arm/Group | Usual Care With LDV/SOF | Usual Care Plus Peer-mentors With LDV/SOF | Usual Care Plus Incentives With LDV/SOF
All-Cause Mortality (participants affected / at risk) | 1/24 | 0/45 | 0/41
Serious Adverse Events (participants affected / at risk) | 3/24 | 9/45 | 9/41
Other Adverse Events (participants affected / at risk) | 11/24 | 18/45 | 19/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care With LDV/SOF (N=24) | Usual Care Plus Peer-mentors With LDV/SOF (N=45) | Usual Care Plus Incentives With LDV/SOF (N=41)
Emphysema/COPD/SOB (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (6)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 6 (6)
Back Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Leg Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2)
Otitis media with effusion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Syncope (General disorders) | 0 (0) | 2 (3) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 2 (3) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Scabies (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Poorly-controlled diabetes (Endocrine disorders) | 0 (0) | 0 (0) | 1 (2)
Hyperkalemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Anion gap metabolic acidosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Decompensated Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Kidney Stones (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Elevated liver enzymes (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Motor Vehicle Accident (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Alcohol withdrawal (Psychiatric disorders) | 0 (0) | 1 (3) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Abcess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
acute congestive heart failure exacerbation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (General disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
cellulitis of left arm during pregnancy (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care With LDV/SOF (N=24) | Usual Care Plus Peer-mentors With LDV/SOF (N=45) | Usual Care Plus Incentives With LDV/SOF (N=41)
Headache (Nervous system disorders) | 5 (6) | 9 (10) | 12 (23)
Fatigue (General disorders) | 6 (7) | 7 (11) | 6 (12)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 3 (10)
Insomnia (General disorders) | 0 (0) | 0 (0) | 6 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes